CLINICAL TRIAL: NCT04281784
Title: Using the Electronic Health Record to Identify and Promote Goals-of-Care Communication for Older Patients With Serious Illness
Brief Title: Project to Improve Communication About Serious Illness--Hospital Study: Pragmatic Trial (Trial 1)
Acronym: PICSI-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, R. Engelberg, Research Professor; Cambia Palliative Care Center of Excellence; Pulmonary, Critical Care and Sleep Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00007031-A; 1R01AG006244 (NIH)
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Dementia; Chronic Disease; Neoplasm Metastasis; Lung Neoplasm; Pulmonary Disease, Chronic Obstructive; Heart Failure，Congestive; Liver Cirrhosis; Kidney Failure, Chronic; Lung Diseases, Interstitial; Peripheral Vascular Disease; Diabetes With End Organ Injury
Keywords: Health care quality, access, and evaluation; Patient care; Inpatients; Health communication; Patient care planning; Palliative care
MeSH Terms: conditions — Dementia; Chronic Disease; Neoplasm Metastasis; Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure; Liver Cirrhosis; Kidney Failure, Chronic; Lung Diseases, Interstitial; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EHR-based Clinician Jumpstart (Experimental): The EHR-based Jumpstart Guide will be developed by extracting data from the EHR using automated methods with both inpatient and outpatient notes (e.g., progress notes, specialty consult notes, alerts and care plans) preceding the current hospitalization. It will summarize the presence/absence of POLST, advance directives and DPOA documentation and patients' code status.
  Interventions: Behavioral: EHR-based Clinician Jumpstart
- Usual Care (No Intervention): The clinicians (hospital teams) for patients in the control group will not receive Jumpstart guides. These subjects will receive usual care.

INTERVENTIONS:
Behavioral: EHR-based Clinician Jumpstart — The Jumpstart Guide is a communication-priming intervention for clinicians that addresses hospitalized patients' goals of care. The intervention's goal is to prompt clinicians to provide standard of care which includes a discussion with patients or their legal surrogate decision-maker about their goals of care. The one-page Jumpstart Guide provides information to the clinician about prior advance care planning documentation and code status derived from the EHR. The Jumpstart Guides includes tips to improve goals-of-care communication.
  Other Names: Jumpstart Guide Intervention; Clinician-facing Jumpstart
  Arms: EHR-based Clinician Jumpstart

SUMMARY:
The objective of this protocol is to test the effectiveness of a Jumpstart intervention on patient-centered outcomes for patients with chronic illness by ensuring that they receive care that is concordant with their goals over time, and across settings and providers. This study will examine the effect of the EHR-based intervention to improve quality of palliative care for patients 55 years or older with chronic, life-limiting illness with a particular emphasis on Alzheimer's disease and related dementias (ADRD). The specific aims are:

1. To evaluate the effectiveness of a novel EHR-based (electronic health record) clinician Jumpstart guide, compared with usual care, for improving the quality of care; the primary outcome is documentation of a goals-of-care discussion in the period between randomization and 30 days following randomization. Secondary outcomes focus on intensity of care: ICU use, ICU and hospital length of stay, costs of care during the hospitalization, and 7 and 30-day hospital readmissions.
2. To conduct a mixed-methods evaluation of the implementation of the intervention, guided by the RE-AIM framework for implementation science, incorporating quantitative evaluation of the intervention's reach and adoption, as well as qualitative analyses of interviews with participants, to explore barriers and facilitators to future implementation and dissemination.

DETAILED DESCRIPTION:
OVERVIEW: This is a large pragmatic trial of the Jumpstart intervention designed to promote goals-of-care discussions for older, seriously ill, hospitalized patients. The trial recruits consecutively eligible patients from three UW Medicine hospitals. The Jumpstart Guide is a communication-priming intervention that addresses hospitalized patients' goals of care. It includes information, drawn from the electronic health record (EHR), identifying the dates and locations of prior advance care planning documents (e.g. living wills, healthcare directives, durable power of attorney for healthcare, and Physician Orders for Life Sustaining Treatments (POLST)) and patients' code status. This information is provided by email to patients' clinicians. The Jumpstart Guide includes tips to improve this communication. The trial will assess the effectiveness of the EHR-based clinician Jumpstart as compared with usual care.

This current study is "Trial 1" of the R01 Award funding this trial. Trial 2 was initiated following the completion of recruitment for Trial 1.

SPECIFIC AIM 1 (for Trial 1): Evaluate the efficacy of the EHR-based clinician Jumpstart compared to usual care for improving quality of care.

TRIAL 1 has three components.

Component 1- Subject Identification/Recruitment/Randomization: The investigators will use automated methods with EHR data, including natural language processing/machine learning (NLP/ML) approaches, to identify hospitalized patients with serious illness during the first 2-3 days of this specific admission. Screening reports will be produced daily and include all likely eligible patients. Study staff will use these daily screening reports to review individual records of eligible patients for inclusion and exclusion criteria (i.e. verify eligibility). Patients will not be approached for consent. Eligible patients will be assigned to intervention or comparator in a 1:1 ratio. Patients are randomized using variable size blocks and stratified for hospital and ADRD vs. no ADRD.

Component 2- EHR-based Clinician Jumpstart Guide: The Jumpstart guide is developed by applying NLP/ML algorithms to both inpatient and outpatient EHR notes (e.g., progress notes, specialty consult notes, alerts and care plans) preceding the current hospitalization. It summarizes the presence/absence of POLST, advance directives and DPOA (durable power of attorney) documentation and the patients' code status. It also provides general recommendations to initiating goals of care discussions. Jumpstart guides are prepared for the intervention group only.

Component 3- Delivery of the intervention: For the intervention group, the investigators deliver the Jumpstart guide to the primary hospital team (attending and resident physicians and advanced practice providers) via secure email. The Jumpstart guides are delivered within 1 business day of patient randomization. Study staff monitor the care team of the patient, and if there are any changes, ensure that any new providers receive the Jumpstart guide as well.

Comparator: The hospital teams for patients in the control group do not receive Jumpstart guides.

Outcome Assessment. Outcomes are obtained from the EHR and use, in part, NLP/ML methods. The primary outcome is EHR documentation of goals-of-care discussions in the 30 days following randomization. Secondary outcomes are measures of intensity of care, including utilization metrics (i.e., ICU admissions, ICU and hospital lengths of stay, 30-day hospital readmissions), costs of care during hospital admission, and estimated costs of implementing the intervention.

SPECIFIC AIM 2 (Trial 1): Evaluate implementation of the Jumpstart Guide and identify barriers and facilitators to future implementation.

Qualitative evaluation:

Clinician recruitment: Study staff will recruit clinicians who were involved with the study to participate in a short interview after the clinician's study involvement with the enrolled patient has ended. Clinician participants will be selected using purposive sampling to ensure a diverse group (e.g., age, race/ethnicity, gender, specialty, year of training).

Interview: Using an interview guide developed specifically for this project, interviewers will assess respondents' experience with the intervention and gather suggestions for ways to improve the intervention's content, delivery and implementation, including implementation outcomes (e.g., acceptability, fidelity, penetration, maintenance) that will guide future dissemination of the intervention.

Assessment: Interviews are audio recorded, transcribed, and analyzed using thematic analytic methods.

Quantitative evaluation:

Quantitative evaluation for Specific Aim 2 will be guided by the RE-AIM framework. We will evaluate the intervention's: 1) Reach (% of all identified eligible clinicians, patients and families that participated in the study); 2) Adoption (% of eligible services that participated); and 3) Implementation (the proportion of HTML Jumpstart Guides that were opened by a clinician, proportion of patients for whom an HTML JS guide was sent and for whom a JS was opened by a clinician).

ELIGIBILITY:
Eligibility criteria apply to two subject groups: 1) seriously ill adult patients; 2) hospital clinicians.

Inclusion Criteria:

* PATIENTS. Eligible patients will be those who are: 1) older than 80 years of age; or 2) 55 years of age or older who meet criteria for serious illness. Serious illness encompasses acute illness (e.g. COVID-19) and chronic illnesses (e.g. those included in the Dartmouth Atlas to study end-of-life care: malignant cancer/leukemia, chronic pulmonary disease, coronary artery disease, heart failure, chronic liver disease, chronic renal disease, dementia, diabetes with end-organ damage, and peripheral vascular disease).
* CLINICIANS (Interview). Eligible clinicians will be those who are 18 years of age or older, English-speaking, employed at a participating hospital, and have been the clinician of record for an enrolled patient in the trial.

Exclusion Criteria:

* Reasons for exclusion for any patient include: restricted status (prisoners or victims of violence); legal or risk management concerns (as determined by the attending physician or via hospital record designation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2512 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Engelberg, PHD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Harborview Medical Center, Seattle, Washington
  - UW Medical Center - Northwest, Seattle, Washington
  - UW Medical Center - Montlake (UWMC), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curtis JR, Lee RY, Brumback LC, Kross EK, Downey L, Torrence J, Heywood J, LeDuc N, Mallon Andrews K, Im J, Weiner BJ, Khandelwal N, Abedini NC, Engelberg RA. Improving communication about goals of care for hospitalized patients with serious illness: Study protocol for two complementary randomized trials. Contemp Clin Trials. 2022 Sep;120:106879. doi: 10.1016/j.cct.2022.106879. Epub 2022 Aug 10. PMID 35963531
- [Result] Curtis JR, Lee RY, Brumback LC, Kross EK, Downey L, Torrence J, LeDuc N, Mallon Andrews K, Im J, Heywood J, Brown CE, Sibley J, Lober WB, Cohen T, Weiner BJ, Khandelwal N, Abedini NC, Engelberg RA. Intervention to Promote Communication About Goals of Care for Hospitalized Patients With Serious Illness: A Randomized Clinical Trial. JAMA. 2023 Jun 20;329(23):2028-2037. doi: 10.1001/jama.2023.8812. PMID 37210665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PATIENTS recruited from 4/23/20 to 3/26/21. A waiver of informed consent and HIPAA authorization obtained for screening and enrollment.
Pre-assignment Details: 4567 potentially eligible patients identified; 4395 patients screened (1883 ineligible, 2512 eligible); 2512 enrolled.
Groups:
- EHR-based Clinician Jumpstart: The EHR-based Jumpstart Guide will be developed by extracting data from the EHR to identify documents uploaded prior to the current hospitalization. It will summarize the presence/absence of POLST, advance directives and DPOA documentation and patients' code status.
  EHR-based Clinician Jumpstart: The Jumpstart Guide is a communication-priming intervention for clinicians that addresses hospitalized patients' goals of care. The intervention's goal is to prompt clinicians to provide standard of care which includes a discussion with patients or their legal surrogate decision-maker about their goals of care. The one-page Jumpstart Guide provides information to the clinician about prior advance care planning documentation and code status derived from the EHR. The Jumpstart Guides includes tips to improve goals-of-care communication.
Period: Overall Study
Arm/Group | EHR-based Clinician Jumpstart | Usual Care
Started | 1255 | 1257
Completed | 1255 | 1257
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EHR-based Clinician Jumpstart | Usual Care | Total
Number analyzed (Participants) | 1255 | 1257 | 2512
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 377 | 412 | 789
  >=65 years | 878 | 845 | 1723
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (10.7) | 71.6 (10.9) | 71.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 543 | 513 | 1056
  Male | 712 | 744 | 1456
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 73 | 150
  Not Hispanic or Latino | 1171 | 1176 | 2347
  Unknown or Not Reported | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 21 | 24 | 45
  Asian | 143 | 149 | 292
  Native Hawaiian or Other Pacific Islander | 4 | 9 | 13
  Black or African American | 168 | 148 | 316
  White | 882 | 886 | 1768
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 37 | 41 | 78
Region of Enrollment [Number; unit: participants]
  United States | 1255 | 1257 | 2512

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With EHR Documentation of Goals of Care Discussions
Description: The primary outcome is the proportion of patients who have a goals-of-care (GOC) discussion that has been documented in the EHR in the period between randomization and 30 days following randomization The proportion is the number of patients with GOC documentation over the number of patients in each study arm. Documentation of goals-of-care discussions will be evaluated using our NLP/ML methods.
Time Frame: Assessed for the period between randomization and 30 days following randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Clinician Jumpstart | Usual Care
Number analyzed (Participants) | 1255 | 1257
Participants
  GOC documented | 433 | 382
  GOC not documented | 822 | 875
Statistical Analysis 1: Comparison: EHR-based Clinician Jumpstart vs Usual Care; Usual care = reference group; intervention arm = comparison group; Test type: Superiority; p = 0.027, Regression, Linear — two-sided test, no adjustment for multiple comparisons; Occurrence of discussion regressed on randomization condition, adjusted for ADRD status, hospital, and time between study start & randomization date; Risk Difference (RD) = 0.0421, 95% CI 2-sided [0.0047 to 0.0777] — Robust standard error

2. Secondary Outcome: Intensity of Care/ICU Use: ICU Admissions
Description: Secondary outcomes include measures of intensity of care, including utilization metrics: Number of ICU admissions during the patient's (index) hospital stay will be collected from the EHR.
Time Frame: Assessed for the period between randomization and 30 days following randomization
Reporting Status: Not Posted

3. Secondary Outcome: Intensity of Care/ICU Use: ICU Length of Stay (Number of Days Alive and Out of the ICU)
Description: Secondary outcomes include measures of intensity of care, including utilization metrics: Number of days alive and out of the ICU within 30 days from randomization will be collected from the EHR.
Time Frame: Assessed for the period between randomization and 30 days following randomization
Measure: Mean (Standard Deviation); unit: days
Groups:
- Usual Care: Patients who received usual care
- EHR-based Clinician Jumpstart: Patients whose care team received the Jumpstart Guide
Arm/Group | Usual Care | EHR-based Clinician Jumpstart
Number analyzed (Participants) | 1257 | 1255
days | 27.90 (6.12) | 27.83 (6.19)
Statistical Analysis 1: Comparison: EHR-based Clinician Jumpstart; Superior outcome for Group 2; Test type: Superiority; p = 0.750, Regression, Linear; Outcome (days alive and out of ICU) regressed on Arm/Group (0=usual care, 1=intervention), adjusted for hospital and ADRD status; Mean Difference (Final Values) = -0.078, 95% CI 2-sided [-0.560 to 0.404], Standard Error of Mean 0.246 — Robust (HC3) standard error

4. Secondary Outcome: Intensity of Care/Hospital Use: Hospital Length of Stay (Number of Days Alive and Out of the Hospital)
Description: Secondary outcomes include measures of intensity of care, including utilization metrics: Number of days alive and out of the hospital within 30 days from randomization will be collected from the EHR.
Time Frame: Assessed for the period between randomization and 30 days following randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care | EHR-based Clinician Jumpstart
Number analyzed (Participants) | 1257 | 1255
days | 21.99 (8.78) | 21.63 (9.15)
Statistical Analysis 1: Comparison: EHR-based Clinician Jumpstart; Superior outcome for Group 2; Test type: Superiority; p = 0.312, Regression, Linear; Outcome (days alive and out of hospital) regressed on Arm/Group (0=usual care, 1=intervention), adjusted for hospital and ADRD status; Median Difference (Final Values) = -0.361, 95% CI 2-sided [-1.060 to 0.338], Standard Error of Mean 0.357 — Robust (HC3) standard error

5. Secondary Outcome: Intensity of Care: Hospital Readmissions 30 Days
Description: Secondary outcomes include measures of intensity of care, including utilization metrics: Proportion of patients readmitted to the hospital following index hospitalization.
Time Frame: Assessed for the period between randomization and 30 days following randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Clinician Jumpstart | Usual Care
Number analyzed (Participants) | 1255 | 1257
Participants | 265 | 251
Statistical Analysis 1: Comparison: EHR-based Clinician Jumpstart vs Usual Care; Usual care = reference group; intervention arm = comparison group; Test type: Superiority; p = 0.475, Regression, Linear — two-sided test, no adjustment for multiple comparisons; Readmission (0, 1) regressed on randomization condition (0=usual care, 1=intervention), adjusted for ADRD status, and hospital site; Risk Difference (RD) = 0.012, 95% CI 2-sided [-0.020 to 0.043] — Robust standard error

6. Secondary Outcome: Intensity of Care: ICU Admissions 30 Days
Description: Secondary outcomes include measures of intensity of care, including utilization metrics: Proportion of patients who received ICU care.
Time Frame: Assessed for the period between randomization and 30 days following randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Clinician Jumpstart | Usual Care
Number analyzed (Participants) | 1255 | 1257
Participants | 336 | 348
Statistical Analysis 1: Comparison: EHR-based Clinician Jumpstart vs Usual Care; Usual care = reference group; intervention arm = comparison group; Test type: Superiority; p = 0.610, Regression, Linear — two-sided test, no adjustment for multiple comparisons; ICU care (0,1) regressed on randomization condition (0=usual care, 1=intervention), adjusted for ADRD status, and hospital site; Risk Difference (RD) = -0.009, 95% CI 2-sided [-0.043 to 0.025] — Robust standard error

7. Secondary Outcome: Total Hospitalization Costs, Randomization to 30 Days After Randomization
Description: Secondary outcomes include measures of intensity of care, including costs of inpatient care, collected from UW Medicine Finance Office and adjusted for inflation.
Time Frame: Assessed for the period between randomization and 30 days later
Population: (Data unavailable from Finance Office for two patients.)
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Usual Care | EHR-based Clinician Jumpstart
Number analyzed (Participants) | 1257 | 1253
US dollars | 21,908.67 (33,613.11) | 22,386.40 (32,988.48)
Statistical Analysis 1: Comparison: EHR-based Clinician Jumpstart; Superior outcome for Group 2; Test type: Superiority — Higher cost indicates worse outcome. Missing if cost data unavailable from Finance Office; p = 0.710, other type of regression; Generalized linear model (gamma family, log link); Outcome on study arm (0=control, 1=intervention) adjusted for hospital and ADRD status, robust SEs; Slope = 0.022, 95% CI 2-sided [-0.092 to 0.135], Standard Error of Mean 0.058 — Robust standard error

8. Secondary Outcome: All-cause Mortality at 30 Days After Randomization (Safety Outcome)
Description: From Washington State death certificates
Time Frame: 30 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | EHR-based Clinician Jumpstart
Number analyzed (Participants) | 1257 | 1255
Participants
  Deceased at 30 days | 64 | 70
  Alive at 30 days | 1193 | 1185
Statistical Analysis 1: Comparison: EHR-based Clinician Jumpstart; Usual care=reference group; intervention arm = comparison group; Test type: Superiority; p = 0.588, Regression, Linear — two-sided test, no adjustment for multiple comparisons; Died within 30 days after randomization regressed on randomization condition (0=usual care, 1=intervention) adjusted for hospital and ADRD status; Risk Difference (RD) = 0.487, 95% CI 2-sided [-1.275 to 2.249], Standard Error of Mean 0.899 — Robust standard error

9. Secondary Outcome: Total Hospitalization Costs, Randomization to Index Hospitalization Discharge
Description: Secondary outcomes include measures of intensity of care, including costs of inpatient care, collected from UW Medicine Finance Office and adjusted for inflation. Assessed for the period between randomization and discharge for the index hospital stay.
Time Frame: Index hospital stay
Population: (Data unavailable from Finance Office for two patients.)
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Usual Care | EHR-based Clinician Jumpstart
Number analyzed (Participants) | 1257 | 1253
US dollars | 24,384.68 (46,677.43) | 23,724.06 (38,623.82)
Statistical Analysis 1: Comparison: EHR-based Clinician Jumpstart; Superior outcome for Group 2; Test type: Superiority — Higher cost indicates worse outcome. Missing if cost data unavailable from Finance Office; p = 0.685, other type of regression; [statistical method as in outcome 7, analysis 1]; Slope = -0.028, 95% CI 2-sided [-0.162 to 0.107], Standard Error of Mean 0.069 — Robust standard error

ADVERSE EVENTS:
Time Frame: Randomization through one year following randomization.
Description: No study-related Serious Adverse Events are expected. The Jumpstart intervention is a communication intervention and is unlikely to result in fatal or life-threatening outcomes.
Arm/Group | EHR-based Clinician Jumpstart | Usual Care
All-Cause Mortality (participants affected / at risk) | 70/1255 | 64/1257
Serious Adverse Events (participants affected / at risk) | 0/1255 | 0/1257
Other Adverse Events (participants affected / at risk) | 0/1255 | 0/1257

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT04281784/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT04281784/SAP_001.pdf